CLINICAL TRIAL: NCT06952595
Title: Carer Involvement in Exercise Programmes for Acute Neurosciences Patients With Acquired Brain Injury
Brief Title: Carer Involvement in Exercises for People With Acquired Brain Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other); 3 Million Steps charity (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 334551 (196-10-23)
Record Dates: First submitted 2025-04-02; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: Stoke; Acquired brain injury; rehabilitation; exercise therapy
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercises for people with acquired brain injury (Experimental)
  Interventions: Behavioral: five exercises prescribed and taught to carers and participants

INTERVENTIONS:
Behavioral: five exercises prescribed and taught to carers and participants — Up to five exercises prescribed and taught to carers and participants in an acute hospital setting fort hem to continue to practice as able.

SUMMARY:
Increasing the amount of exercises completed has been shown to help recovery for people after a brain injury. This study will explore if providing extra training of exercises prescribed to a patient and carer team, will allow more practice of these exercises, better abilities to move and balance, and to assess if carer confidence changes with doing this. It is a repeated case design in the in-patient acute Neurosciences setting at the Norfolk and Norwich University Hospital NHS Trust (NNUH).

ELIGIBILITY:
Inclusion

* Adults with acquired brain injury on NNUH Neurosciences Unit with a carer physically able to complete exercises with the patient.
* Patient to be able to follow simple commands (1 stage) for exercise intervention.
* Patient able to consent along with their relative together to participation in the study.

Exclusion:

* Discharge plan for ESD from initial assessment with no care package required due to too short timeframe of being an acute in-patient.
* Patient's with severe cognitive - communication deficits meaning they cannot follow 1 stage command for exercises or consent to the study.
* Severe pain, joint abnormality or spasticity limiting participation in exercise programme.
* Carer/relative not able to physically help the patient with the required exercises or carer/relative not able to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Log of exercise repetitions | Pre and post intervention: 4 weeks or at point of discharge from acute Trust.
  Log of exercise repetitions completed by patient and relative/carer team (on exercise record log), VAS score (Visual analogue score) rating 0- no confidence to 10- very confident for carer confidence pre and post intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, United Kingdom